CLINICAL TRIAL: NCT02636023
Title: A Clinical Study to Determine the Correlation Between the SPhENo-Cardiograph™, a Seismocardiograph Device, and GE Vivid Q, an Echocardiograph, for Known Systemic Timing Intervals (STI).
Brief Title: Correlation Between the SPhENo-Cardiograph™, a Seismocardiograph Device, and GE Vivid Q, an Echocardiograph, for Known Systemic Timing Intervals (STI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Force Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SPHENO_CLIN_003
Record Dates: First submitted 2015-10-22; First posted 2015-12-21 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPhENo-Cardiograph / ECG (Experimental): SPhENo-Cardiograph and ECG
  Interventions: Device: SPhENo-Cardiograph

INTERVENTIONS:
Device: SPhENo-Cardiograph — SPhENo-Cardiograph

SUMMARY:
The study Sponsor, Heart Force Medical Inc. (HFM), has developed a patented medical device called the SPhENo-CardiographTM. The SPhENo-Cardiograph™ provides a non-invasive assessment of the electro-mechanical function of the heart. The electrocardiograph (ECG) represents the waveform of the electrical stimulus to the cardiac muscle. The mechanical actions of the electrical potentials delivered in the ECG are revealed as the seismocardiograph (SCG). The SCG represents the changes in acceleration of the heart during the cardiac cycle. The SCG waveform reflects the ultra-low frequency vibrations of cardiac contraction. These low frequency vibrations are transmitted through the sternum. Using the point of initiation of ventricular contraction on the ECG, the Q wave, with fiduciary points on the synchronous seismocardiograph, it is possible to determine timing events of the cardiac cycle. The timing events of the cardiac cycle during systole are referred to as Systolic Timing Intervals (STI) and comprise the Pre-Ejection Period (PEP) and the Left Ventricular Ejection Time (LVET). The PEP is the time from the Q wave to the Aortic valve opening. The Left Ventricular Eject Time (LVET) is the time between the Aortic Valve opening and closing. The ratio of PEP/LVET in individuals with established heart disease is > 0.42. It is based on the formula described by Dr Arnold Weissler and first published in Circulation in 1968 (Weissler et al,1968). Weissler et al showed that the PEP/LVET ratio >0.42 are indicative of a lengthening of the PEP with some marginal shortening of the LVET. This is indicative of pathology associated with the coronary circulation (Ahmed et al, 1972;). This ratio can then be used as part of a non-invasive quantitative assessment of cardiac performance (Lewis et al 1977).

Using the SPhENo-CardiographTM, HFM has developed an algorithm to assess heart health that otherwise requires a number of technologies; stethoscope, ECG and Carotid pulse tracing to identify the dicrotic notch or Aortic Valve closure.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the informed consent document
* Willing to participate in study
* Ambulatory volunteer

Exclusion Criteria:

* Individuals with visible scar(s) or deformity in the test area of the chest
* Non-ambulatory subjects
* Previously diagnosed with life-threatening condition (e.g. cancer)
* Known or diagnosed psychiatric condition
* Enrolled in a concurrent study or trial
* Exercised excessively within the last 4 hours (prior to study visit)
* Consumption of caffeine containing drinks within the previous 4 hours
* Unwilling to sign Informed Consent
* Female subjects who are pregnant, suspected or planning to become pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient ≥0.8 between STI ratio values determined by the SPhENo-Cardiograph™ and an echocardiograph | 1 day
Correlation coefficient ≥0.8 between PEP values determined by the SPhENo-Cardiograph™ and an echocardiograph | 1 day
Correlation coefficient ≥0.8 between LVET values determined by the SPhENo-Cardiograph™ and an echocardiograph | 1 day
Correlation coefficient ≥0.8 between heart rate values determined by the SPhENo-Cardiograph™ and an echocardiograph | 1 day

SECONDARY OUTCOMES:
Correlation coefficient ≥0.8 between STI ratio values determined by the SPhENo-Cardiograph™ and a manual analysis | 1 day
Correlation coefficient ≥0.8 between PEP values determined by the SPhENo-Cardiograph™ and a manual analysis | 1 day
Correlation coefficient ≥0.8 between LVET values determined by the SPhENo-Cardiograph™ and a manual analysis | 1 day
Correlation coefficient ≥0.8 between heart rate values determined by the SPhENo-Cardiograph™ and a manual analysis | 1 day
Safety and tolerability assessed by Adverse event collection | 1 day
  Adverse event collection
Subject questionnaire | 1 day
  Questionnaire to evaluate relevance of device from subject's perspective; data to be analyzed qualitatively

CONTACTS AND LOCATIONS:
Overall Officials: Karrin Fairman Young, ND, Principal Investigator — Boucher Institute of Naturopathic Medicine
Locations (1):
- Boucher Institute of Naturopathic Medicine, New Westminster, British Columbia, Canada